CLINICAL TRIAL: NCT04705142
Title: Beneficial Effect of Intravenous Magnesium Sulphate in Term Neonates With Hypoxic Ischemic Encephalopathy(HIE)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Services Institute of Medical Sciences, Pakistan (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ref No. IRB/2019/527/SIMS
Record Dates: First submitted 2020-11-21; First posted 2021-01-12 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: HIE
Keywords: HIE, MgSO4

STUDY DESIGN:
Intervention Model Description: Case control study
Masking Description: Blinded Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MgSO4 (Experimental): MgSO4
  1st dose within 6 hours of life @250mg/kg,2nd after 24 hours of life @250mg/kg, 3rd after 48 hours of life @250mg/kg.
  Monitoring and Protective measures:
  Before and during administration of MgSO4, B.P, Capillary refill time, Heart rate and respiratory rate will be assessed closely i-e on 10 minutes interval, infusion of MgSO4 will be give over 30 minutes and baby will be monitored every 15 minutes interval after completion of infusion as well for 1 hour.
  Interventions: Drug: MgSo4

INTERVENTIONS:
Drug: MgSo4 — Before and during administration of MgSO4, B.P, Capillary refill time, Heart rate and respiratory rate will be assessed closely i-e on 10 minutes interval, infusion of MgSO4 will be give over 30 minutes and baby will be monitored every 15 minutes interval after completion of infusion as well for 1 hour.
  Other Names: Conventional Treatment

SUMMARY:
Neonatal mortality rate is the highest in Pakistan. And Birth Asphyxia is one of the main reversible causes. Outcomes related to birth asphyxia can be improved, if intervention done in time with proper measures. MgSO4 is cheaper and easily available drug.

DETAILED DESCRIPTION:
Some studies showed positive results if given within 6 hours of birth asphyxia, whereas some are not supportive. But still less know about this drug, especially in low income countries. Objective of this study is to see beneficial effects of MgSO4 in neonates presenting with birth asphyxia.

ELIGIBILITY:
Inclusion Criteria:

* After informed consent, any child who is term, inborn or out born fulfilling the definition of hypoxic ischemic encephalopathy according to history, apgar or scoring system and reaching within 6 hours of delivery in nursery department of pediatric medicine unit-II, Services Hospital, Lahore

Exclusion Criteria:

* Preterm Syndromic/dysmorphic child Term child with HIE and arriving after 6 hours of life. Term child with unrelated co morbidities eg congenital heart defects, Renal failure etc

Max Age: 6 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Reduction in Immediate complications of disease | 2 weeks
  Reduction in Immediate complications of disease
Reduction in mortality | 2 weeks
  Reduction in mortality
Reduction in hospital stay | 2 weeks
  Reduction in hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Dr Uzair Ahmed, MBBS, FCPS, Study Director — Associate Prof, Surgery
Locations (1):
- Services Institute of Medical Sciences, Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
After family consent, decision will be reviewed

REFERENCES:
- [Background] Gathwala G, Khera A, Singh J, Balhara B. Magnesium for neuroprotection in birth asphyxia. J Pediatr Neurosci. 2010 Jul;5(2):102-4. doi: 10.4103/1817-1745.76094. PMID 21559152
- See also: Reference Study — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3087983/